CLINICAL TRIAL: NCT02357485
Title: Adipose Derived Stromal Cell (ADSC) Injections for Pain Management of Osteoarthritis in the Human Knee Joint
Brief Title: ADSC Injections for Pain Management of Osteoarthritis in the Human Knee Joint
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fodor, Peter B, M.D. (Individual)
Collaborators: Plastic Surgery Education and Research Foundation (Unknown)
Responsible Party: Principal Investigator, Peter B. Fodor MD, Peter B. Fodor, M.D., Fodor, Peter B, M.D.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OAKnee01
Record Dates: First submitted 2015-01-31; First posted 2015-02-06 (Estimated); Results first posted 2015-03-27 (Estimated); Last update posted 2015-06-30 (Estimated); Status verified 2015-06

CONDITIONS: Osteoarthritis of the Knee
Keywords: ADSC; osteoarthritis; knee; adipose
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment arm (Experimental): Single injection of ADSC
  Interventions: Biological: ADSC

INTERVENTIONS:
Biological: ADSC — Single injection of ADSC

SUMMARY:
This safety and feasibility study used autologous adipose-derived stromal cells (ADSC), the stromal vascular fraction (SVF), to treat 8 osteoarthritic (OA) knees in 6 patients of grade I to III (K-L scale) with initial pain of 4 or greater on a 10 point scale, under Institutional Review Board (IRB) approved protocol.

DETAILED DESCRIPTION:
This safety and feasibility study used autologous adipose-derived stromal cells, the stromal vascular fraction, to treat 8 osteoarthritic knees in 6 patients of grade I to III (K-L scale) with initial pain of 4 or greater on a 10 point scale, under IRB-approved protocol. Evaluation of the safety of intra-articular injection of the stromal vascular fraction cells was the primary objective of the study. Adipose-derived stromal vascular cells were obtained through enzymatic disaggregation of lipoaspirate, resuspended in 3 ml of Lactated Ringer's Solution, and injected directly into the intra-articular space with a mean of 12 million viable nucleated SVF cells per knee.

ELIGIBILITY:
Inclusion Criteria:

* voluntarily provided written Informed Consent
* ages 20-70
* male or female
* grades I-III radiologically documented OA of one or both knees
* American Society Anaesthesiologists (ASA) physical status class I-II and a • BMI less than 35
* knee pain graded as greater than 3 out of 10 on screening questionnaire
* able to speak, read and understand English -

Exclusion Criteria:

* patient parameters falling outside of the inclusion criteria
* current oral or parenteral steroid or blood thinner use
* hyaluronic acid-based injection to the affected knee joint within the previous six months
* corticosteroid injection to the affected knee joint within the previous three months
* end stage (Grade IV) OA

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-03; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter B Fodor, M.D., Principal Investigator — Private Practice

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Arm: Single injection of Adipose-derived Stromal Cells (ADSC) into intra-articular space of the knee
Period: Overall Study
Arm/Group | Treatment Arm
Started | 6 (6 subjects, 8 knees ( 2 bilateral & 4 unilateral))
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Six (6) participants with eight (8) knees - Two (2) participants with bilateral OA (4 knees) Four (4) participant with unilateral OA (4 knees)
Arm/Group | Treatment Arm
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.3 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 1

OUTCOME MEASURES:

1. Primary Outcome: Safety as Measured by Adverse Events
Description: Adverse Events were recorded during the entirety of the study.
Time Frame: Entire Study (1 year)
Population: All 6 participants were included in the analysis
Measure: Number; unit: percentage of participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 6
percentage of participants | 0

2. Secondary Outcome: Comparison of Baseline Score and 1 Year Score in Western Ontario and McMaster Universities Arthritis Index (WOMAC)
Description: Comparison of WOMAC score (pain, stiffness and functionality measures) measured at baseline (pre-treatment), 3 months and 1 year (post treatment).
  WOMAC score: 0 (best) to 100 (worst)
Time Frame: Baseline to 1 year
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: knees
Arm/Group | Treatment Arm
Number analyzed (Participants) | 6
Number analyzed (knees) | 8
units on a scale
  Pre-treatment | 32.9 (14.6)
  3 months Post-treatment | 10.8 (13.1)
  1 year Post-treatment | 9.3 (11.4)
Statistical Analysis 1: Comparison: Treatment Arm; Test type: Superiority or Other; p < 0.004, t-test, 2 sided — Baseline vs 1 year Post-treatment

3. Secondary Outcome: Comparison of Baseline Score and 1 Year Score in Visual Analog Scale (VAS) for Pain
Description: Comparison of VAS pain score as measured before treatment and 3 months and 1 year after treatment. VAS measured on a scale of 0 (no pain) to 10 (worst possible pain).
Time Frame: Baseline to 1 year
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: knees
Arm/Group | Treatment Arm
Number analyzed (Participants) | 6
Number analyzed (knees) | 8
units on a scale
  Pre-treatment | 5.9 (1.2)
  3 months Post-treatment | 1.8 (2.6)
  1 year Post-treatment | 2.0 (2.0)
Statistical Analysis 1: Comparison: Treatment Arm; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — Baseline vs 1 year Post-treatment

4. Secondary Outcome: Comparison of Baseline and 3 Months Measures of Knee Flexion for Range of Motion
Description: Comparison of baseline measure of knee flexion to 3 months measurements of knee flexion. An increase in range of motion is positive (improved ability to move) and a decrease in range of motion is negative.
Time Frame: Baseline to 3 months
Measure: Mean (Standard Deviation); unit: degrees
Units Other Than Participants: knees
Arm/Group | Treatment Arm
Number analyzed (Participants) | 6
Number analyzed (knees) | 8
degrees
  Pre-treatment | 136.6 (7.3)
  Post-treatment | 143.6 (6.7)
Statistical Analysis 1: Comparison: Treatment Arm; Test type: Superiority or Other; p = 0.053, t-test, 2 sided

5. Secondary Outcome: Comparison of Baseline Score and 3 Months Score in Timed-Up-and-Go (TUG).
Description: Comparison of baseline time for subjects' ability to rapidly rise from a chair, move rapidly 2 meters from the chair, turn and return and sit in the chair to the same measure at 3 months. Time to complete task is measured in seconds.
Time Frame: baseline to 3 months
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Treatment Arm
Number analyzed (Participants) | 6
seconds
  Pre-treatment | 5.4 (1.6)
  Post-treatment | 2.8 (0.3)
Statistical Analysis 1: Comparison: Treatment Arm; Test type: Superiority or Other; p = 0.003, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Treatment Arm
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No